CLINICAL TRIAL: NCT07216326
Title: Our Voices Matter: Racial Justice Activism Intervention to Address Structural Racism and Prevent Depression in Black and Latinx Youth
Brief Title: Our Voices Matter: Intervention for Depression in Youth
Acronym: OVM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Policy Research Associates (Unknown)
Responsible Party: Principal Investigator, Nia Heard-Garris, Assistant Professor of Pediatrics, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB 2024-6683; 1R01MD017610-01A1 (NIH)
Record Dates: First submitted 2024-12-09; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Depressive Symptoms; Allostatic Load; Metabolic Syndrome
Keywords: mental health; youth intervention; allostatic load; stress; depressive symptoms; depression; metabolic syndrome; prevention; inflammation
MeSH Terms: conditions — Depression; Metabolic Syndrome; Psychological Well-Being; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RJA Intervention Arm (Experimental): The "Our Voices Matter" RJA intervention is a block-stratified randomized, group behavioral intervention designed for Black and Latinx adolescents and young adults (AYAs). The curriculum will specifically focus on the principles of education, organizing, policy development, and legal advocacy. Participants will have didactic sessions, which include policy debates, keynote lectures, seminars, and trainings led by local leaders, community activists, and other experts on civil rights. Participants will learn how to use data to understand how structural barriers influence life. Participants will understand and analyze policy and develop action plans to influence SRD. Additionally, the program will create a network of supportive peers. After the RJA training, small groups will meet monthly via videoconference for 1-year post-intervention. This intervention aims to equip Black and Latinx AYAs with civic and grassroots organizing knowledge and peer support.
  Interventions: Behavioral: Racial Justice Activism Intervention ARM
- Adulting 101 (Placebo Comparator): Adulting 101: Life Skills attention control is a 5- day in-person program that will meet for the same number of sessions and duration as the intervention. This attention control is based on the "Project Life" program developed initially for individuals supporting youth transitioning out of foster care to teach life skills for independent living. This curriculum is delivered through didactic and interactive modules that provide knowledge and informational resources, along with hands-on activities and life skills demonstrations. Sessions include: 1) Community Building, 2) Career Preparation, 3) Education, 4) Money Management, 5) Health and Nutrition, 6) Home Management, and 7) Story Sharing.
  Interventions: Behavioral: Adulting 101- Control Arm

INTERVENTIONS:
Behavioral: Racial Justice Activism Intervention ARM — The "Our Voices Matter" RJA intervention is a block-stratified randomized, group behavioral intervention designed for Black and Latinx adolescents and young adults (AYAs). The curriculum will specifically focus on the principles of activism, organizing, policy development, and legal advocacy. Participants will have didactic sessions, which include policy debates, keynote lectures, seminars, and trainings led by local leaders, community activists, and other experts on civil rights. Participants will learn how to use data to understand how structural racism and discrimination (SRD) influence life. Participants will understand and analyze policy and develop action plans to influence SRD. Additionally, the program will create a network of supportive peers. After the RJA training, small groups will meet monthly via videoconference for 1-year post-intervention. This intervention aims to equip Black and Latinx AYAs with civic and grassroots organizing knowledge and peer support.
  Other Names: RJA Intervention ARM
  Arms: RJA Intervention Arm
Behavioral: Adulting 101- Control Arm — Adulting 101: Life Skills attention control is a 5- day in-person program (Figure 4) that will meet for the same number of sessions and duration as the intervention. This attention control is based on the "Project Life" program,84 developed initially for individuals supporting youth transitioning out of foster care to teach life skills for independent living. This curriculum is delivered through didactic and interactive modules that provide knowledge and informational resources, along with hands-on activities and life skills demonstrations. Sessions include: 1) Community Building, 2) Career Preparation, 3) Education, 4) Money Management, 5) Health and Nutrition, 6) Home Management, and 7) Story Sharing, which culminates with a Day of Action. Participants will learn skills for adulthood and gain experience developing career and education goals. Like the intervention condition, participants will actualize their skills on the final day, called the "Day of Action."
  Other Names: Adulting/RJA Control
  Arms: Adulting 101

SUMMARY:
Over 15 million people participated in racial justice protests nationwide during 2020-2021 spotlighting activism as a collective tool against structural racism and discrimination (SRD). SRD manifests as policies and practices (e.g., redlining, voter suppression, mass incarceration) that produce hostile environments that contribute to psychological distress, elevated allostatic load, and an elevated risk for chronic diseases and premature death, concentrated within Black and Latinx populations. While the connection between SRD and health is well documented, few studies provide evidence on strategies to reduce SRD and mitigate consequences on psychological and physiological outcomes. Thus, there is a critical need to rigorously test interventions that improve the mental and physical health of Black and Latinx populations, beginning in adolescence. The study's specific aims are to 1) Determine whether a racial justice activism behavioral intervention prevents and reduces depressive symptoms in Black and Latinx adolescents and young adults and 2) Determine whether a racial justice activism behavioral intervention lowers allostatic load scores in Black and Latinx adolescents and young adults. To accomplish these aims, the team will conduct a stage II group-based, multi-component, and multilevel randomized behavioral clinical trial. The investigators will collect psychological and physiological measures at baseline, then at defined intervals for 2 years post the racial justice activism intervention.

DETAILED DESCRIPTION:
The investigators will conduct a phase II group-based, multi-component, and multi-level randomized behavioral clinical trial. The investigators will recruit and enroll 300 participants aged 15-20 (N=150 intervention and N=150 control) in Chicago, Illinois. After enrollment, participants will be randomized using a block-stratified randomization technique to ensure balance regarding race, ethnicity, and gender. Once participants are recruited, the investigators will use a computer-generated random number sequence to assign participants to the intervention group (Racial Justice Activism) or control group (Adulting 101: Life Skills Training). Participants assigned to the intervention arm will participate in 5 half-day interactive sessions teaching grassroots organizing and activism specific to SRD. Participants will be assigned to the control arm and will participate in 5 half-day interactive sessions teaching life skills training. Following the activism training, the intervention arm participants will meet virtually in small peer groups to continue advocacy for group-identified SRD issues. Following the life skill attention control programs, control arm participants will meet virtually in small peer groups to continue refresher and discussion of life skills. Participants in the control arm will undergo life skills training with the same number of sessions and duration as the intervention arm.

Participants in both the intervention and control arms will report depressive symptoms on a clinically relevant measure (e.g., Patient Health Questionnaire-9) at baseline and then <1-, 6-, 12-, 18-, and 24- months post-initial 5-day activism or life skills training. In addition to depressive symptoms, the investigators will measure other aspects of psychological distress, including anxiety and stress as secondary outcomes. Participants in both groups will have biometric samples, like blood draws, and clinical measurements of allostatic load at baseline and then 6-,12-, and 24- months post-initial 5-day activism or life skills training.

The proposed project will use a cluster randomized trial that involves complete groups of individuals randomized to conditions (i.e., intervention, control), with clustering occurring in both arms. All of our statistical analyses will appropriately model the dependency among observations, which is a hallmark of multi-level modeling.

ELIGIBILITY:
Inclusion Criteria:

1. 15-20 years old
2. Identify as Black and/ or Latinx
3. Speak English

Exclusion Criteria:

1. Younger than 15 years old, or older than 20 years old
2. Unable to attend the in-person sessions
3. Non-fluent English speaker
4. Do not identify as Black or Latinx

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptoms | at baseline and then 0-1-, 6-, 12-, 18-, and 24- months post initial 5 day-intervention
  To evaluate depressive symptoms and overall depression, the investigators will use the following measurement tools: the Patient Questionnaire-9 [PHQ-9]. The investigators have chosen these metrics because these tools have been validated within our study population and the PHQ-9 is used in clinical practice. The Patient Health Questionnaire-9 (PHQ-9) is used in clinical practice to diagnose and manage depression and has a minimal clinically important difference (MCID) of 5 points on the PHQ-9 total score. The minimum is a score of 0 and the maximum is a score of 27, with higher scores indicating worse depressive symptoms. The scoring is as follows: Scores 0-4: None/minimal depression, 5-9: mild depression, 10-14: moderate depression, 15-19: moderately severe depression, 20-27: severe depression.
Metabolic Syndrome | at baseline and then 6-, 12-, and 24- months post initial 5 day-intervention
  Biomarkers will be collected from these systems: cardiovascular (e.g., systolic and diastolic blood pressure (measured in mmHg), serum triglycerides (mg/dL) and HDL cholesterol (mg/dL), metabolic (e.g., glycosylated hemoglobin [HbA1c-(mg/dL)] , fasting glucose (mg/dL), waist circumference (cm), and insulin (U/ML).
  Will measure seated blood pressure, height (cm), weight (Kg), and waist circumference using the same protocols used in the HCHS/SOL Youth for rigor and reproducibility.
  To arrive at one reported value of metabolic syndrome, we will
  1. a count of the number of signs that meet International Diabetes Federation (IDF) criteria, and
  2. also create continuous metabolic risk score. To calculate this score, each biomarker will have values standardized into a z-score, then sum the z-scores, (Before transformation waist circumference will be normed for age, sex, and race using nationally representative data from NHANES.)
Blood Pressure | at baseline and then 6-, 12-, and 24- months post initial 5 day-intervention
  The investigators will measure systolic and diastolic blood pressure (measured in mmHg) using a size-appropriate blood pressure cuff.
Triglycerides | at baseline and then 6-, 12-, and 24- months post initial 5 day-intervention
  The investigators will measure serum triglycerides (mg/dL) as a component of lipid markers.
High-density lipoprotein | at baseline and then 6-, 12-, and 24- months post initial 5 day-intervention
  The investigators will measure HDL cholesterol (mg/dL) as a component of lipid markers.
Glycosylated hemoglobin | at baseline and then 6-, 12-, and 24- months post initial 5 day-intervention
  The investigators will measure HbA1c (mg/dL) as a marker of metabolic health.
Glucose | at baseline and then 6-, 12-, and 24- months post initial 5 day-intervention
  The investigators will measure fasting glucose (mg/dL) as a marker of metabolic health.
Insulin | at baseline and then 6-, 12-, and 24- months post initial 5 day-intervention
  The investigators will measure insulin (U/ML) as a marker of metabolic health.
Waist Circumference | at baseline and then 6-, 12-, and 24- months post initial 5 day-intervention
  The investigators will measure waist circumference (cm) as a marker of metabolic health.

SECONDARY OUTCOMES:
Perceived Stress | at baseline and then 0-1 month, 6-, 12-, 18-, and 24- months post initial 5 day-intervention
  The investigators will use the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Short Form on psychological stress experiences to enhance rigor and reproducibility. This tool has acceptable reliability and validity in AYAs. The scoring range is 4-20, with higher scores indicating greater stress severity.
Anxiety | at baseline and then 0-1 month, 6-, 12-, 18-, and 24- months post initial 5 day-intervention
  Anxiety will be measured using the Generalized Anxiety Disorder Questionnaire-7 (GAD-7). The GAD-7 has been validated with our study population and is used in clinical practice with an MCID of 4 points on the GAD-7 total score. The scoring is as follows: 0-4: Minimal anxiety, 5-9: Mild anxiety,10-14: Moderate anxiety, and 15-21: Severe anxiety.
Inflammation | at baseline and then 6-, 12-, and 24- months post initial 5 day-intervention
  The investigators will use biomarkers from inflammatory/immune systems (e.g., Hs-CRP (mg/L), IL-1β (pg/mL), IL-6 (pg/mL), IL-8 (pg/mL), suPAR (pg/mL), and TNF-α (pg/mL). The investigators plan to measure an inflammation score, by standardizing values each biomarker into a z-score, then sum the z-scores to arrive at one reported inflammation score.
C-Reactive Protein | at baseline and then 6-, 12-, and 24- months post initial 5 day-intervention
  The investigators will measure Hs-CRP (mg/L) as a measure of inflammation.
Interleukin-1βeta | at baseline and then 6-, 12-, and 24- months post initial 5 day-intervention
  The investigators will measure IL-1β (pg/mL) as measure of inflammation.
Interleukin-6 | at baseline and then 6-, 12-, and 24- months post initial 5 day-intervention
  The investigators will measure IL-6 (pg/mL) as a measure of inflammation.
Interleukin-8 | at baseline and then 6-, 12-, and 24- months post initial 5 day-intervention
  The investigators will measure IL-8 (pg/mL) as a measure of inflammation.
Soluble Urokinase Plasminogen Activator Receptor (suPAR) | at baseline and then 6-, 12-, and 24- months post initial 5 day-intervention
  The investigators will measure suPAR (pg/mL) as a measure of inflammation.
Tumor Necrosis Factor alpha (TNF-α) | at baseline and then 6-, 12-, and 24- months post initial 5 day-intervention
  The investigators will measure TNF-α (pg/mL) as a measure of inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Elan C Hope, PhD, Principal Investigator — Policy Research Associates
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Northwestern Univ. (NU) and Lurie Children's (LCH) are committed to the open and timely dissemination of all research outcomes through the development of repositories and databases, posting of data on open websites, presentations, and through publications as soon as is feasible after peer review. Team will assure the confidentiality of all human subjects' data and will adhere to all HIPAA rules to ensure compliance with human subject confidentiality requirements. Collaborators will ensure that any data obtained as a part of the awarded grant will be made available to collaborators and to the general research community through databases and public repositories and by publishing in printed or electronic form as soon as practically possible after the data have been obtained and peer-reviewed. Team agrees to publish all data derived from this award in a timely fashion and to make those data freely available via web postings whenever possible. All data will be made available after 1 year.
Supporting Information: Study Protocol
Time Frame: Research data will be made publicly available through posting on open websites, presentations, and peer-reviewed publications (in some cases after an embargo period not to exceed one year). Inventions appropriate for commercialization will be protected via intellectual property (IP) filings, commercialized, and provided to society as products or services by or through the Innovation and New Ventures Office, NU's technology transfer office. Innovation and New Ventures Office manages NU's invention disclosure, assessment, patenting, and marketing processes. NU is committed to the free exchange of data and resources and for the rapid commercialization of biomedical inventions for the benefit of the public, consistent with the terms of the Bayh-Dole Act. NU's commercialization practices to date have maximized the public benefit of inventions arising from federal funding by providing useful, commercially relevant, and available products and services.
Access Criteria: Data and resource sharing is an essential to the study activities. The team will share the data and resources generated by this project by making our findings, intervention materials and protocols (e.g., training materials, manuals, etc.), available to the following communities:
  1. Scientists interested in developing, implementing, and testing activism as an approach to reduce the health risks associated with structural racism, particularly among adolescent and young adult populations. Data and resource sharing with this community will encourage dialogue about the nuances of activism as a youth health intervention, implementation, and evaluation research in youth-focused community settings.
  2. Practitioners, clinicians, youth educators, administrators, and other decision-makers, so our findings may be used to inform youth civic education and advocacy programming;
  3. The community at large, so adolescents, young adults, and their caregivers and educators can use our findings

REFERENCES:
- [Background] Pinedo A, Durkee MI, Diemer MA, Hope EC. Disentangling longitudinal trajectories of racial discrimination and critical action among Black and Latinx college students: What role do peers play? Cultur Divers Ethnic Minor Psychol. 2021 Jul;27(3):546-557. doi: 10.1037/cdp0000434. Epub 2021 Apr 29. PMID 33914581
- [Background] Volpe VV, Schorpp KM, Cacace SC, Benson GP, Banos NC. State- and Provider-Level Racism and Health Care in the U.S. Am J Prev Med. 2021 Sep;61(3):338-347. doi: 10.1016/j.amepre.2021.03.008. Epub 2021 Jun 24. PMID 34419231
- [Background] Gaydosh L, Schorpp KM, Chen E, Miller GE, Harris KM. College completion predicts lower depression but higher metabolic syndrome among disadvantaged minorities in young adulthood. Proc Natl Acad Sci U S A. 2018 Jan 2;115(1):109-114. doi: 10.1073/pnas.1714616114. Epub 2017 Dec 18. PMID 29255040
- [Background] Volpe VV, Lee DB, Hoggard LS, Rahal D. Racial Discrimination and Acute Physiological Responses Among Black Young Adults: The Role of Racial Identity. J Adolesc Health. 2019 Feb;64(2):179-185. doi: 10.1016/j.jadohealth.2018.09.004. Epub 2018 Nov 6. PMID 30409752
- [Background] Hope EC, Brinkman M, Hoggard LS, Stokes MN, Hatton V, Volpe VV, Elliot E. Black adolescents' anticipatory stress responses to multilevel racism: The role of racial identity. Am J Orthopsychiatry. 2021;91(4):487-498. doi: 10.1037/ort0000547. Epub 2021 Apr 22. PMID 34338546
- [Background] Cohen A, Ekwueme PO, Sacotte KA, Bajwa L, Gilpin S, Heard-Garris N. "Melanincholy": A Qualitative Exploration of Youth Media Use, Vicarious Racism, and Perceptions of Health. J Adolesc Health. 2021 Aug;69(2):288-293. doi: 10.1016/j.jadohealth.2020.12.128. Epub 2021 Feb 19. PMID 33612361
- [Background] Ballard PJ, Syme SL. Engaging youth in communities: a framework for promoting adolescent and community health. J Epidemiol Community Health. 2016 Feb;70(2):202-6. doi: 10.1136/jech-2015-206110. Epub 2015 Oct 6. PMID 26443541
- [Background] Heard-Garris N, Ekwueme PO, Gilpin S, Sacotte KA, Perez-Cardona L, Wong M, Cohen A. Adolescents' Experiences, Emotions, and Coping Strategies Associated With Exposure to Media-Based Vicarious Racism. JAMA Netw Open. 2021 Jun 1;4(6):e2113522. doi: 10.1001/jamanetworkopen.2021.13522. PMID 34129023
- [Background] Hope EC, Velez G, Offidani-Bertrand C, Keels M, Durkee MI. Political activism and mental health among Black and Latinx college students. Cultur Divers Ethnic Minor Psychol. 2018 Jan;24(1):26-39. doi: 10.1037/cdp0000144. Epub 2017 Jun 26. PMID 28650179
- [Background] Banales J, Aldana A, Richards-Schuster K, Flanagan CA, Diemer MA, Rowley SJ. Youth anti-racism action: Contributions of youth perceptions of school racial messages and critical consciousness. J Community Psychol. 2021 Nov;49(8):3079-3100. doi: 10.1002/jcop.22266. Epub 2019 Nov 6. PMID 31691984
- [Background] Lee DB, Peckins MK, Heinze JE, Miller AL, Assari S, Zimmerman MA. Psychological pathways from racial discrimination to cortisol in African American males and females. J Behav Med. 2018 Apr;41(2):208-220. doi: 10.1007/s10865-017-9887-2. Epub 2017 Sep 23. PMID 28942527
- [Background] Hill LK, Hoggard LS, Richmond AS, Gray DL, Williams DP, Thayer JF. Examining the association between perceived discrimination and heart rate variability in African Americans. Cultur Divers Ethnic Minor Psychol. 2017 Jan;23(1):5-14. doi: 10.1037/cdp0000076. PMID 28045306
- [Background] Chae DH, Nuru-Jeter AM, Adler NE, Brody GH, Lin J, Blackburn EH, Epel ES. Discrimination, racial bias, and telomere length in African-American men. Am J Prev Med. 2014 Feb;46(2):103-11. doi: 10.1016/j.amepre.2013.10.020. PMID 24439343
- [Background] Adam EK, Heissel JA, Zeiders KH, Richeson JA, Ross EC, Ehrlich KB, Levy DJ, Kemeny M, Brodish AB, Malanchuk O, Peck SC, Fuller-Rowell TE, Eccles JS. Developmental histories of perceived racial discrimination and diurnal cortisol profiles in adulthood: A 20-year prospective study. Psychoneuroendocrinology. 2015 Dec;62:279-91. doi: 10.1016/j.psyneuen.2015.08.018. Epub 2015 Aug 28. PMID 26352481
- [Background] Hicken MT, Lee H, Ailshire J, Burgard SA, Williams DR. "Every shut eye, ain't sleep": The role of racism-related vigilance in racial/ethnic disparities in sleep difficulty. Race Soc Probl. 2013 Jun 1;5(2):100-112. doi: 10.1007/s12552-013-9095-9. PMID 23894254
- [Background] Turan B, Foltz C, Cavanagh JF, Wallace BA, Cullen M, Rosenberg EL, Jennings PA, Ekman P, Kemeny ME. Anticipatory sensitization to repeated stressors: the role of initial cortisol reactivity and meditation/emotion skills training. Psychoneuroendocrinology. 2015 Feb;52:229-38. doi: 10.1016/j.psyneuen.2014.11.014. Epub 2014 Nov 22. PMID 25497480
- [Background] Alegria M, Shrout PE, Canino G, Alvarez K, Wang Y, Bird H, Markle SL, Ramos-Olazagasti M, Rivera DV, Cook BL, Musa GJ, Falgas-Bague I, NeMoyer A, Dominique G, Duarte C. The effect of minority status and social context on the development of depression and anxiety: a longitudinal study of Puerto Rican descent youth. World Psychiatry. 2019 Oct;18(3):298-307. doi: 10.1002/wps.20671. PMID 31496076
- [Background] Assari S, Moazen-Zadeh E, Caldwell CH, Zimmerman MA. Racial Discrimination during Adolescence Predicts Mental Health Deterioration in Adulthood: Gender Differences among Blacks. Front Public Health. 2017 May 29;5:104. doi: 10.3389/fpubh.2017.00104. eCollection 2017. PMID 28611972
- [Background] Perreira KM, Marchante AN, Schwartz SJ, Isasi CR, Carnethon MR, Corliss HL, Kaplan RC, Santisteban DA, Vidot DC, Van Horn L, Delamater AM. Stress and Resilience: Key Correlates of Mental Health and Substance Use in the Hispanic Community Health Study of Latino Youth. J Immigr Minor Health. 2019 Feb;21(1):4-13. doi: 10.1007/s10903-018-0724-7. PMID 29550906
- [Background] Cardoso JB, Szlyk HS, Goldbach J, Swank P, Zvolensky MJ. General and Ethnic-Biased Bullying Among Latino Students: Exploring Risks of Depression, Suicidal Ideation, and Substance Use. J Immigr Minor Health. 2018 Aug;20(4):816-822. doi: 10.1007/s10903-017-0593-5. PMID 28493116
- [Background] Nguyen-Rodriguez ST, Gallo LC, Isasi CR, Buxton OM, Thomas KS, Sotres-Alvarez D, Redline S, Castaneda SF, Carnethon MR, Daviglus ML, Perreira KM. Adiposity, Depression Symptoms and Inflammation in Hispanic/Latino Youth: Results From HCHS/SOL Youth. Ann Behav Med. 2020 Jun 12;54(7):529-534. doi: 10.1093/abm/kaz070. PMID 32043152
- [Background] Utsey, S. O., Belvet, B., Hubbard, R. R., Fischer, N. L., Opare-Henaku, A., & Gladney, L. L. (2013). Development and validation of the Prolonged Activation and Anticipatory Race-Related Stress Scale. Journal of Black Psychology, 39(6), 532-559.
- [Background] Brody GH, Lei MK, Chae DH, Yu T, Kogan SM, Beach SRH. Perceived discrimination among African American adolescents and allostatic load: a longitudinal analysis with buffering effects. Child Dev. 2014 May-Jun;85(3):989-1002. doi: 10.1111/cdev.12213. Epub 2014 Feb 5. PMID 24673162
- [Background] Paradies Y, Ben J, Denson N, Elias A, Priest N, Pieterse A, Gupta A, Kelaher M, Gee G. Racism as a Determinant of Health: A Systematic Review and Meta-Analysis. PLoS One. 2015 Sep 23;10(9):e0138511. doi: 10.1371/journal.pone.0138511. eCollection 2015. PMID 26398658
- [Background] Ong AD, Williams DR, Nwizu U, Gruenewald TL. Everyday unfair treatment and multisystem biological dysregulation in African American adults. Cultur Divers Ethnic Minor Psychol. 2017 Jan;23(1):27-35. doi: 10.1037/cdp0000087. PMID 28045308
- [Background] Lockwood KG, Marsland AL, Matthews KA, Gianaros PJ. Perceived discrimination and cardiovascular health disparities: a multisystem review and health neuroscience perspective. Ann N Y Acad Sci. 2018 Sep;1428(1):170-207. doi: 10.1111/nyas.13939. Epub 2018 Aug 8. PMID 30088665
- [Background] Lewis TT, Cogburn CD, Williams DR. Self-reported experiences of discrimination and health: scientific advances, ongoing controversies, and emerging issues. Annu Rev Clin Psychol. 2015;11:407-40. doi: 10.1146/annurev-clinpsy-032814-112728. Epub 2015 Jan 2. PMID 25581238
- [Background] Hope EC, Kornbluh M, Hagan M, Davis AL, Alexander A. Validation of the Black Community Activism Orientation Scale with racially and ethnically diverse college students. Am J Community Psychol. 2023 Mar;71(1-2):79-89. doi: 10.1002/ajcp.12633. Epub 2022 Nov 15. PMID 36378747
- [Background] Hope EC, Gugwor R, Riddick KN, Pender KN. Engaged Against the Machine: Institutional and Cultural Racial Discrimination and Racial Identity as Predictors of Activism Orientation among Black Youth. Am J Community Psychol. 2019 Mar;63(1-2):61-72. doi: 10.1002/ajcp.12303. Epub 2019 Jan 18. PMID 30659621
- [Background] Hope EC, Cryer-Coupet QR, Stokes MN. Race-related stress, racial identity, and activism among young Black men: A person-centered approach. Dev Psychol. 2020 Aug;56(8):1484-1495. doi: 10.1037/dev0000836. PMID 32790447